CLINICAL TRIAL: NCT01180504
Title: Consolidation Intensity-Modulated Whole Abdominal Radiotherapy for High-Risk Patients With Ovarian Cancer Stage FIGO III
Brief Title: Consolidation Whole Abdominal Intensity-Modulated Radiation Therapy (IMRT) in Advanced Ovarian Cancer
Acronym: OVAR-IMRT-02
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Juergen Debus / Prof., M.D., PhD, Department of Radiation Oncology, University of Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVAR-IMRT-02
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Ovarian Cancer; Tubal Carcinoma; Primary Peritoneal Carcinoma
Keywords: ovarian cancer; whole-abdominal radiotherapy; consolidation treatment; helical tomotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: intensity-modulated whole-abdominal radiotherapy — Consolidation intensity-modulated whole-abdominal radiotherapy using helical tomotherapy to a total dose of 30 Gy in 1.5 Gy fractions

SUMMARY:
The primary objective of this phase-II study is to assess the toxicity of consolidation intensity-modulated whole-abdominal radiotherapy using tomotherapy in patients with advanced optimally debulked stage International Federation of Gynecology and Obstetrics (FIGO) III ovarian cancer with a complete remission after adjuvant chemotherapy.

36 patients will be treated to a total dose of 30 Gy in 1.5 Gy fractions. The planning target-volume includes the entire peritoneal cavity and the pelvic and para-aortal node regions. Intensity-modulated whole-abdominal radiotherapy allows an effective sparing of liver, kidneys and bone-marrow (vertebral bodies and pelvic bones).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed ovarian cancer or tube cancer or primary peritoneal carcinoma stage FIGO III
* primary optimal debulking surgery
* postoperative gross residual tumor ≤ 1cm ( R0, R1 oder R2 < 1cm situation)
* adjuvant chemotherapy with platin and taxane
* complete remission after chemotherapy
* Karnofsky performance score > 60
* patients >18 years of age
* written informed consent

Exclusion Criteria:

* stage FIGO I or II
* stage III with postoperative gross residual tumor > 1cm
* stage FIGO IV
* recurrence situation
* delayed wound healing post laparotomy
* leucopenia <2000/ml before radiotherapy
* thrombocytopenia <75000/ml before radiotherapy
* clinically active renal, hepatic, cardiac, metabolic, respiratory, coagulation or hematopoietic disease
* status post pelvic or abdominal radiotherapy
* status post other cancer disease in the past 5 years (cervical cancer in situ, basal cell carcinoma, squamous cell carcinoma of the skin are excluded)
* participation in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
compatibility of the treatment | Beginning of radiotherapy till 6 weeks after its completion
  Therapy compatibility defined as non-occurrence of life-threatening grade 4 (CTCAE v3.0) acute toxicity

SECONDARY OUTCOMES:
Rate of incomplete radiotherapy | 4 weeks
  Rate of incomplete radiotherapy due to treatment toxicity
Rate of delayed radiotherapy | 4 weeks
  Rate of delayed radiotherapy due to treatment toxicity
Acute toxicity | From the beginning of radiotherapy till 6 weeks after its completion
  Graded according CTCAE Version 3.0
Late Toxicity | 6 weeks -3 years after the completion of radiotherapy
  Graded according CTCAE Version 3.0
Overall survival | 3 years
Disease-free survival | 3 years after the completion of radiotherapy
Quality of life | 3 years
  assessed using EORTC QLQ-C30 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schneeweiss, MD, Principal Investigator — Department of Gyneacology and Obstetrics, Unversity of Heidelberg; Juergen Debus, MD, PhD, Principal Investigator — Department of Radiation Oncology, University of Heidelberg
Locations (1):
- Department of Radiation Oncology, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Rochet N, Sterzing F, Jensen AD, Dinkel J, Herfarth KK, Schubert K, Eichbaum MH, Schneeweiss A, Sohn C, Debus J, Harms W. Intensity-modulated whole abdominal radiotherapy after surgery and carboplatin/taxane chemotherapy for advanced ovarian cancer: phase I study. Int J Radiat Oncol Biol Phys. 2010 Apr;76(5):1382-9. doi: 10.1016/j.ijrobp.2009.03.061. Epub 2009 Jul 21. PMID 19628341
- [Derived] Arians N, Kieser M, Benner L, Rochet N, Schroder L, Katayama S, Herfarth K, Schubert K, Schneeweiss A, Sohn C, Lindel K, Debus J. Adjuvant intensity modulated whole-abdominal radiation therapy for high-risk patients with ovarian cancer FIGO stage III: final results of a prospective phase 2 study. Radiat Oncol. 2019 Oct 21;14(1):179. doi: 10.1186/s13014-019-1381-2. PMID 31639066
- [Derived] Rochet N, Kieser M, Sterzing F, Krause S, Lindel K, Harms W, Eichbaum MH, Schneeweiss A, Sohn C, Debus J. Phase II study evaluating consolidation whole abdominal intensity-modulated radiotherapy (IMRT) in patients with advanced ovarian cancer stage FIGO III--the OVAR-IMRT-02 Study. BMC Cancer. 2011 Jan 28;11:41. doi: 10.1186/1471-2407-11-41. PMID 21276234